CLINICAL TRIAL: NCT07070739
Title: A Multicenter, Open-label Study to Evaluate the Long-term Safety and Efficacy of HSK44459 Tablets for the Treatment of Patients With Bechet's Disease
Brief Title: A Long-term Study of HSK44459 Tablets in Participants With Bechet's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK44459-205
Record Dates: First submitted 2025-07-09; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Bechet's Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: HSK44459 tablets

INTERVENTIONS:
Drug: HSK44459 tablets — Orally, twice a day

SUMMARY:
This is a long-term extension study of HSK44459-202 in eligible participants who have completed the Week 12 visit of the originating Study HSK44459-202. The total duration of this study will be up to 56 weeks which will include a 52-week treatment period, and a 4-week safety follow-up period after the last study intervention administration. Safety will be assessed by the incidence and severity of adverse events during the study.

ELIGIBILITY:
Inclusion Criteria:

- Have previously participated in clinical studies on the treatment of Bechet's disease with HSK44459 tablets and completed the specified treatment in accordance with the protocol;

Exclusion Criteria:

1. Active involvement of major organs related to Behçet's disease - pulmonary (eg, pulmonary artery aneurysms), vascular (eg, thrombophlebitis), gastrointestinal (eg, gastrointestinal ulcers), and central nervous system (eg, meningoencephalitis) manifestations, and ocular lesions (eg, uveitis) requiring immunosuppressive treatment.
2. Subjects who experienced treatment-emergent serious adverse events (SAEs) related to the investigational product in previous HSK44459 studies, and in the investigator's judgment, are not suitable for continuing treatment with HSK44459 tablets.
3. Currently has hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or has other clinically active liver disease, or tests positive for HBsAg or anti-HCV
4. Subjects whom the investigator deems to have any other factors that make them unsuitable for participating in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events during the study | 56 weeks

SECONDARY OUTCOMES:
Complete remission rate of oral ulcers | 52 weeks
Changes in oral ulcer pain measured by VAS compared with baseline | 52 weeks
Changes in Bechet's Disease Quality of Life Score (BD-QoL) compared with baseline | 52 weeks
Changes in the Short Form Health Survey (SF-36) compared with baseline | 52 weeks